CLINICAL TRIAL: NCT04362670
Title: A Randomized, Multi-center, Double-masked, Vehicle-controlled, Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of OTX-CSI (Cyclosporine Ophthalmic Insert) for Intracanalicular Use for the Treatment of Subjects With Dry Eye Disease (DED)
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of OTX-CSI in Subjects With Dry Eye Disease.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CLN-Protocol-0054
Record Dates: First submitted 2020-04-16; First posted 2020-04-27 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Dry Eye Disease
Keywords: Cyclosporine; Intracanalicular insert
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Sequential: Groups of participants are assigned to receive interventions based on prior milestones being reached in the study, such as in some dose escalation and adaptive design studies
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- OTX-CSI-Cohort 1 (Experimental): Formulation 2A-.36 mg
  Interventions: Drug: OTX-CSI
- OTX-CSI-Cohort 2 (Experimental): Formulation 1- .36 mg
  Interventions: Drug: OTX-CSI
- HV (Placebo Comparator): Cohort 2:
  Formulation 2B
  Interventions: Other: Placebo Vehicle
- OTX-CSI- Cohort 2 (Experimental): Formulation 2A- .36 mg
  Interventions: Drug: OTX-CSI
- HV-2 (Placebo Comparator): Cohort 2:
  Formulation 3
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: OTX-CSI — OTX-CSI intracanalicular insert
  Arms: OTX-CSI- Cohort 2; OTX-CSI-Cohort 1; OTX-CSI-Cohort 2
Other: Placebo Vehicle — Hydrogel Vehicle intracanalicular insert
  Arms: HV; HV-2

SUMMARY:
To assess the safety, tolerability and efficacy of a single dose of OTX-CSI, a sustained release cyclosporine drug product, in subjects with dry eye disease.

DETAILED DESCRIPTION:
Randomized, multi-center, double-masked, vehicle-controlled, Phase 1/2 study to evaluate the safety, tolerability, and efficacy of OTX-CSI in subjects with dry eye disease. The subjects will be followed for approximately 16 weeks after product insertion

ELIGIBILITY:
Inclusion Criteria:

* Dry eye disease diagnosis
* VAS eye dryness severity score ≥ 30.

Exclusion Criteria:

* Are unwilling to discontinue use of contact lenses
* Are unwilling to withhold use of artificial tears.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Ocular Therapeutix, Inc., Garden Grove, California
  - Ocular Therapeutix, Inc., Inglewood, California
  - Ocular Therapeutix, Inc., Mission Hills, California
  - Ocular Therapeutix, Inc., Delray Beach, Florida
  - Ocular Therapeutix, Inc., Largo, Florida
  - Ocular Therapeutix, Inc., Lake Villa, Illinois
  - Ocular Therapeutix, Inc., Kansas City, Missouri
  - Ocular Therapeutix, Inc, St Louis, Missouri
  - Ocular Therapeutix, St Louis, Missouri
  - Ocular Therapeutix, Inc., Cleveland, Ohio
  - Ocular Therapeutix, Inc., Cranberry Township, Pennsylvania
  - Ocular Therapeutix, Inc., Memphis, Tennessee
  - Ocular Therapeutix, Inc., El Paso, Texas
  - Ocular Therapeutix, Lakeway, Texas
  - Ocular Therapeutix, Inc., Murray, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- OTX-CSI Cohort 1 F2A: This arm was open label and all 5 subjects received F2A OTX-CSI 0.36 mg Cyclosporine Ophthalmic Insert (expected approximate persistence 3-4 months)
- OTX-CSI Cohort 2 F1: Subjects in this arm received OTX-CSI 0.36 mg Cyclosporine Ophthalmic Insert (expected approximate persistence 2-3 months)
- OTX-CSI Cohort 2 F2A: Subjects in this arm received OTX-CSI 0.36 mg Cyclosporine Ophthalmic Insert (expected approximate persistence 3-4 months)
- OTX-CSI Cohort 2 F2B: Subjects in this arm received Hydrogel Vehicle Insert (expected approximate persistence 3-4 months)
- OTX-CSI Cohort 2 F3: Subjects in this arm received Hydrogel Vehicle Insert (expected approximate persistence 1 week)
Period: Overall Study
Arm/Group | OTX-CSI Cohort 1 F2A | OTX-CSI Cohort 2 F1 | OTX-CSI Cohort 2 F2A | OTX-CSI Cohort 2 F2B | OTX-CSI Cohort 2 F3
Started | 5 | 42 | 41 | 43 | 22
Completed | 5 | 39 | 39 | 42 | 22
Not Completed | 0 | 3 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-CSI Cohort 1 F2A | OTX-CSI Cohort 2 F1 | OTX-CSI Cohort 2 F2A | OTX-CSI Cohort 2 F2B | OTX-CSI Cohort 2 F3 | Total
Number analyzed (Participants) | 5 | 42 | 41 | 43 | 22 | 153
Age, Categorical [Count of Participants; unit: Participants] — Population: Cohort 1 and the Modified Intent-to-Treat (mITT) population (defined as all subjects who received the insert in the study eye).
  Participants
    number analyzed (Participants) | 5 | 42 | 40 | 43 | 22 | 152
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 1 | 16 | 13 | 19 | 8 | 57
    >=65 years | 4 | 26 | 27 | 24 | 14 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (8.1) | 67.9 (10.2) | 68.0 (11.5) | 65.5 (10.4) | 65.2 (9.7) | 67.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Cohort 1 and the Modified Intent-to-Treat (mITT) population (defined as all subjects who received the insert in the study eye).
  Participants
    number analyzed (Participants) | 5 | 42 | 40 | 43 | 22 | 152
    Female | 5 | 29 | 25 | 39 | 17 | 115
    Male | 0 | 13 | 15 | 4 | 5 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort 1 and the Modified Intent-to-Treat (mITT) population (defined as all subjects who received the insert in the study eye).
  Participants
    number analyzed (Participants) | 5 | 42 | 40 | 43 | 22 | 152
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 6 | 7 | 8 | 2 | 23
    White | 5 | 36 | 33 | 34 | 18 | 126
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Population: Cohort 1 and the Modified Intent-to-Treat (mITT) population (defined as all subjects who received the insert in the study eye).
  participants
    North America: number analyzed (Participants) | 5 | 42 | 40 | 43 | 22 | 152
    North America | 5 | 42 | 40 | 43 | 22 | 152

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With At Least One (1) Treatment Emergent Adverse Event
Description: Number of Subjects With At Least One (1) Treatment Emergent Adverse Event
Time Frame: From Screening to Study Exit, approximately 156 days.
Measure: Number; unit: count of participants
Arm/Group | OTX-CSI Cohort 1 F2A | OTX-CSI Cohort 2 F1 | OTX-CSI Cohort 2 F2A | OTX-CSI Cohort 2 F2B | OTX-CSI Cohort 2 F3
Number analyzed (Participants) | 5 | 42 | 41 | 43 | 22
count of participants | 0 | 16 | 15 | 5 | 1

2. Primary Outcome: Schirmer Test Score, CFB at Week 12
Description: A Schirmer test strip measures the amount of tear production and provides a unit of measure in millimeters (mm).
Time Frame: Change from Baseline at Week 12
Population: Cohort 1 was not included in this analysis, as Cohort 1 was evaluated for Safety only.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | OTX-CSI Cohort 1 F2A | OTX-CSI Cohort 2 F1 | OTX-CSI Cohort 2 F2A | OTX-CSI Cohort 2 F2B | OTX-CSI Cohort 2 F3
Number analyzed (Participants) | 0 | 42 | 40 | 43 | 22
millimeters |  | 1.98 [0.04 to 3.92] | 1.91 [-0.01 to 3.82] | 2.24 [0.38 to 4.10] | 3.08 [0.51 to 5.65]

ADVERSE EVENTS:
Time Frame: approximately 156 days
Description: "OTX-CSI Cohort 2F1","OTX-CSI Cohort 2 F2A", and"OTX-CSI Cohort 2 F2B" Arms had 16, 15, and 5 participants, respectively, who experienced at least 1 Treatment Emergent Adverse Event (TEAE).Of these 16, 15, and 5 participants, some experienced more than 1 TEAE. Since some subjects reported more than 1 TEAE, the count of participants in Section 1 (subjects that reported at least 1 TEAE) may not match the sum of Affected subjects in the "SAE" and the "Other (Not Including Serious) AE" sections
Arm/Group | OTX-CSI Cohort 1 F2A | OTX-CSI Cohort 2 F1 | OTX-CSI Cohort 2 F2A | OTX-CSI Cohort 2 F2B | OTX-CSI Cohort 2 F3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/42 | 0/41 | 0/43 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/42 | 2/41 | 0/43 | 0/22
Other Adverse Events (participants affected / at risk) | 0/5 | 15/42 | 14/41 | 5/43 | 1/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-CSI Cohort 1 F2A (N=5) | OTX-CSI Cohort 2 F1 (N=42) | OTX-CSI Cohort 2 F2A (N=41) | OTX-CSI Cohort 2 F2B (N=43) | OTX-CSI Cohort 2 F3 (N=22)
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
COVID-19 Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-CSI Cohort 1 F2A (N=5) | OTX-CSI Cohort 2 F1 (N=42) | OTX-CSI Cohort 2 F2A (N=41) | OTX-CSI Cohort 2 F2B (N=43) | OTX-CSI Cohort 2 F3 (N=22)
Eye Disorders (Eye disorders) | 0 | 13 | 11 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04362670/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT04362670/SAP_001.pdf